CLINICAL TRIAL: NCT05711758
Title: Efficacy and Safety of Endoscopic Antral Myotomy as a Novel Weight Loss Procedure: A Pilot Study
Brief Title: Efficacy and Safety of Endoscopic Antral Myotomy as a Novel Weight Loss Procedure
Acronym: PSAM
Status: Recruiting | Type: Observational
Sponsor: Christopher C. Thompson, MD, MSc (Other)
Responsible Party: Sponsor-Investigator, Christopher C. Thompson, MD, MSc, Director of Endoscopy, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Other Study IDs: 2022P003420
Record Dates: First submitted 2022-12-29; First posted 2023-02-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Obesity, Morbid; Obesity, Primary; Metabolic Disease; Delayed Gastric Emptying Following Procedure
Keywords: Pylorus Sparing Antral Myotomy (PSAM); Gastric physiology; Gastric emptying; Pylorus-sparing antral myotomy; Myotomy; Endoscopic Sleeve Gastroplasty (ESG); TransPyloric Shuttle (TPS); Intragastric balloon (IGB); Endoscopic bariatric and metabolic therapies (EBMT); Gut Hormones; Gastric Emptying Breath Test
MeSH Terms: conditions — Obesity; Obesity, Morbid; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PSAM Treatment Patients with no prior endoscopic bariatric therapies: Subjects with no prior endoscopic bariatric therapies having esophagogastroduodenoscopy (EGD) with Pylorus Sparing Antral Myotomy (PSAM) with standard of care lifestyle modification therapy.
  Interventions: Procedure: PSAM Treatment Patients
- PSAM Treatment Patients with prior primary endoscopic bariatric therapies: Subjects with prior primary endoscopic bariatric therapies having esophagogastroduodenoscopy (EGD) with Pylorus Sparing Antral Myotomy (PSAM) with standard of care lifestyle modification therapy.
  Interventions: Procedure: PSAM Treatment Patients
- PSAM Treatment Patients with prior revision endoscopic bariatric therapies: Subjects with prior revision endoscopic bariatric therapies having esophagogastroduodenoscopy (EGD) with Pylorus Sparing Antral Myotomy (PSAM) with standard of care lifestyle modification therapy.
  Interventions: Procedure: PSAM Treatment Patients

INTERVENTIONS:
Procedure: PSAM Treatment Patients — PSAM is a pylorus-sparing antral myotomy performed under general anesthesia. Endoscopic myotomy is then performed applying the principles of submucosal endoscopy and techniques used during gastric per-oral endoscopic myotomy (G-POEM). A submucosal bleb is created proximal to the pylorus. A longitudinal mucosal incision is made with an endoscopic knife. The endoscope is then introduced into the submucosal space, and the knife is used to dissect the submucosal fibers. Antral myotomy is performed starting proximal to the pyloric ring extending to the mucosal access site. The myotomy entails cutting of the inner circular and oblique muscle bundles or may be full thickness at the discretion of the endoscopist. The mucosal entry is then closed using endoscopic suturing or clips.
  Other Names: PSAM

SUMMARY:
Gastric myotomy has been performed for several years as a means of addressing chronic stenosis after sleeve gastrectomy and treating gastroparesis. The Pylorus Sparing Antral Myotomy (PSAM) technique has the opposite effect by leaving the pylorus intact and extending the myotomy proximally to the distal gastric body. PSAM was initially combined with ESG and shown to delay gastric emptying and provide greater weight loss without impacting tolerability (GCSI score) or the safety profile of the procedure (2 DDW GEM abstracts). PSAM has not been evaluated alone, without concomitant ESG. Since delayed gastric emptying alone is known to promote weight loss, it is thought that PSAM alone (without ESG) may provide similar efficacy, while reducing procedure time and adverse events. There have been no clinical studies that investigate the efficacy of PSAM independent of ESG. This pilot study aims to address this lack of information by evaluating the safety, tolerability, and short-term efficacy of PSAM, in addition to exploring its impact on gastric physiology. This will also provide data that may be used in designing a larger clinical trial.

DETAILED DESCRIPTION:
Obesity, defined as body mass index (BMI) greater than 30 kg/m2 in adults, is affecting 30% of the global population and a significant healthcare burden. [1] Obesity has increased dramatically over the last few decades, with over 650 million adults, or 13% of the world's total adult population, diagnosed with the disease in 2016 - a figure that has nearly tripled since 1975.[1] In the U.S the obesity prevalence for U.S. adults increased from 14.1% to 26.7%, or an 89.9% increase between 1993 and 2008.[1,2,3] As a result, current and potential interventions, and treatment strategies to combat obesity have become more important.

The current treatment of obesity involves multiple strategies with combination of non-pharmacologic, pharmacologic, endoscopic, and surgical interventions. There are several FDA-approved pharmacotherapies for the treatment of obesity such as orlistat, phentermine-topiramate, naltrexone-bupropion, liraglutide, and semaglutide. For adults with a body mass index (BMI) of 40 kg/m2 or 35 kg/m2 and obesity-related comorbidity, bariatric surgery can be offered. [4, 5] Endoscopic bariatric and metabolic therapies (EBMT) have emerged as an alternative treatment for patients with obesity with a BMI over 30kg/m2 or 27 kg/m2 with an obesity-related comorbidity. The interest in EBMT is growing given their safety, efficacy, and non-invasive nature. Current FDA-cleared devices that can be used for EBMT include intragastric balloons and suturing devices for endoscopic sleeve gastroplasty (ESG). Additionally, a variety of Endo surgical knifes are approved for tissue dissection such as myotomy.

Gastric interventions used to treat obesity work by interfering with gastric accommodation, breakdown and mixing of food, or gastric emptying. Delaying gastric emptying was shown to be a major mechanism of action for both ESG and IGB which is also correlated with weight loss [6].

Antral peristalsis constitutes an important mechanism for gastric emptying. The antrum also serves as a food sensor which needs to be filled to a certain level before food is pumped into the duodenum. [7] Therefore, targeting the antrum is a feasible strategy to delay gastric emptying, induce satiety, and promote weight loss.

In fact, one of the recently FDA-cleared EBMT devices, the Transpyloric Shuttle (Baronova, MA), focuses on inhibiting the antral pump as its primary mechanism of action. This device consists of two interconnected large and small bulbs, positioned in the antrum and duodenum respectively, that cause intermittent obstruction of the pylorus, leading to a delay in gastric emptying (10).

As such, a pylorus sparing antral myotomy (PSAM) with a submucosal tunneling technique was developed. Gastric myotomy has been performed for several years as a means of addressing chronic stenosis after sleeve gastrectomy and treating gastroparesis. The PSAM technique has the opposite effect by leaving the pylorus intact and extending the myotomy proximally to the distal gastric body. PSAM was initially combined with ESG and shown to delay gastric emptying and provide greater weight loss without impacting tolerability (GCSI score) or the safety profile of the procedure (2 DDW GEM abstracts). PSAM has not been evaluated alone, without concomitant ESG. Since delayed gastric emptying alone is known to promote weight loss, it is thought that PSAM alone (without ESG) may provide similar efficacy, while reducing procedure time and adverse events.

Traditional bariatric surgery is very effective at treating obesity, however, only 1% of eligible patients elect to undergo this treatment option. Additionally, the majority of patients with obesity do not qualify for bariatric surgery. [5] Due to the less invasive nature of PSAM, and relative technical simplicity compared to ESG) this procedure may provide a more widely available and more acceptable treatment option for some patients.

There have been no clinical studies that investigate the efficacy of PSAM independent of ESG. This pilot study aims to address this lack of information by evaluating the safety, tolerability, and short-term efficacy of PSAM, in addition to exploring its impact on gastric physiology. This will also provide data that may be used in designing a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* subjects must be 18-70 years of age
* eligible for endoscopic and surgical weight loss procedures
* body mass index (BMI) greater than 35 kg/m2
* Individuals must be in excellent mental health
* able to understand and sign informed consent
* available to return for all routine follow-up study visits

Exclusion Criteria:

* untreated H. pylori infection
* gastroparesis
* active smoking
* an ongoing or a history of treatment with opioids in the last 12 months prior to enrollment
* previous pyloromyotomy or pyloroplasty
* gastrointestinal obstruction
* severe coagulopathy
* esophageal or gastric varices and/or portal hypertensive gastropathy
* pregnancy or puerperium
* any inflammatory disease of the gastrointestinal tract (including but not limited to severe (LA Grade C or D) esophagitis, active gastric ulceration, active duodenal ulceration, or specific inflammation such as Crohn's disease)
* malignant or premalignant gastric diseases (such as high grade dysplasia, gastric cancer, or GIST)
* severe cardiopulmonary disease or a history of coronary artery disease (including myocardial infarction within the past 6 months, poorly controlled hypertension, required use of NSAIDs)
* lactation
* history of gastrointestinal surgery
* any serious health condition unrelated to their weight that would increase the risk of endoscopy
* chronic abdominal pain
* active psychological issues preventing participation in a lifestyle modification program
* a known history of endocrine disorders affecting weight (uncontrolled hypothyroidism)
* an inability to provide informed consent
* use of any medication that may interfere with weight loss
* use of any medication that may interfere with gastric emptying
* any other condition which the investigator may deem as an impediment to compliance or hinder completion of the proposed study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults in the Center for Weight Management and Wellness program at Brigham and Women's Hospital with a BMI >35 kg/m2 who are pre-qualified by their insurance as recommended by their specialist to undergo an endoscopic bariatric procedure.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight change compared to baseline | Screening, Procedure day, 1 month, 3 month, 6 month, 9 month, 12 months
  Percent total body weight loss
Adverse Events | Procedure day, 1 month, 3 month, 6 month, 9 month, 12 months
  Changes to health compared to baseline
Change in tolerability from procedure day to 12 months | Procedure day, 1 month, 3 month, 6 month, 9 month, 12 months
  How the subjects feel after the procedure based on pain scale and AE's

SECONDARY OUTCOMES:
Change in Quality of Life compared to baseline | Screening, 1 month, 3 month, 6 month, 9 month, 12 months
  Overall quality of life questionnaire
Gastric Emptying compared to baseline | Screening, 6 months, 12 months
  Gastric emptying using a gastric emptying breath test (GEBT)
Ghrelin levels compared to baseline | Screening, 6 months, 12 months
  Laboratory analysis of blood samples to test ghrelin levels
Insulin levels compared to baseline | Screening, 6 months, 12 months
  Laboratory analysis of blood samples to test insulin metabolic profiles
HgA1c levels compared to baseline | Screening, 6 months, 12 months
  Laboratory analysis of blood samples to test HgA1c metabolic profiles
Glucose levels compared to baseline | Screening, 6 months, 12 months
  Laboratory analysis of blood samples to test Glucose metabolic profiles
HOMA-IR blood plasma levels compared to baseline | Screening, 6 months, 12 months
  Laboratory analysis of blood samples to test changes in insulin resistance
Physiologic Changes of gastric motility/transit compared to baseline | Screening, 6 months, 12 months
  Upper GI series comparing pre-procedure barium transit to post-procedure 6 and 12 month time points.
Gastric Motility compared to baseline | Screening, 1 month
  Dynamic MRI

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. Thompson, MD, MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study to collect data for a larger NIH grant submission, we do not have plans to share data at this time.

REFERENCES:
- [Background] Klem ML, Wing RR, Chang CC, Lang W, McGuire MT, Sugerman HJ, Hutchison SL, Makovich AL, Hill JO. A case-control study of successful maintenance of a substantial weight loss: individuals who lost weight through surgery versus those who lost weight through non-surgical means. Int J Obes Relat Metab Disord. 2000 May;24(5):573-9. doi: 10.1038/sj.ijo.0801199. PMID 10849578
- [Background] James PT, Leach R, Kalamara E, Shayeghi M. The worldwide obesity epidemic. Obes Res. 2001 Nov;9 Suppl 4:228S-233S. doi: 10.1038/oby.2001.123. PMID 11707546
- [Background] Jia H, Lubetkin EI. Obesity-related quality-adjusted life years lost in the U.S. from 1993 to 2008. Am J Prev Med. 2010 Sep;39(3):220-7. doi: 10.1016/j.amepre.2010.03.026. PMID 20709253
- [Background] Tak YJ, Lee SY. Anti-Obesity Drugs: Long-Term Efficacy and Safety: An Updated Review. World J Mens Health. 2021 Apr;39(2):208-221. doi: 10.5534/wjmh.200010. Epub 2020 Mar 9. PMID 32202085
- [Background] Abu Dayyeh BK, Rajan E, Gostout CJ. Endoscopic sleeve gastroplasty: a potential endoscopic alternative to surgical sleeve gastrectomy for treatment of obesity. Gastrointest Endosc. 2013 Sep;78(3):530-5. doi: 10.1016/j.gie.2013.04.197. Epub 2013 May 24. PMID 23711556
- [Background] Gomez V, Woodman G, Abu Dayyeh BK. Delayed gastric emptying as a proposed mechanism of action during intragastric balloon therapy: Results of a prospective study. Obesity (Silver Spring). 2016 Sep;24(9):1849-53. doi: 10.1002/oby.21555. Epub 2016 Jul 28. PMID 27465076
- [Background] Abu Dayyeh BK, Acosta A, Camilleri M, Mundi MS, Rajan E, Topazian MD, Gostout CJ. Endoscopic Sleeve Gastroplasty Alters Gastric Physiology and Induces Loss of Body Weight in Obese Individuals. Clin Gastroenterol Hepatol. 2017 Jan;15(1):37-43.e1. doi: 10.1016/j.cgh.2015.12.030. Epub 2015 Dec 31. PMID 26748219
- [Background] Goyal RK, Guo Y, Mashimo H. Advances in the physiology of gastric emptying. Neurogastroenterol Motil. 2019 Apr;31(4):e13546. doi: 10.1111/nmo.13546. Epub 2019 Feb 10. PMID 30740834
- [Background] Aghaie Meybodi M, Qumseya BJ, Shakoor D, Lobner K, Vosoughi K, Ichkhanian Y, Khashab MA. Efficacy and feasibility of G-POEM in management of patients with refractory gastroparesis: a systematic review and meta-analysis. Endosc Int Open. 2019 Mar;7(3):E322-E329. doi: 10.1055/a-0812-1458. Epub 2019 Feb 28. PMID 30842971
- [Background] Mohan BP, Chandan S, Jha LK, Khan SR, Kotagiri R, Kassab LL, Ravikumar NPG, Bhogal N, Chandan OC, Bhat I, Hewlett AT, Jacques J, Ponnada S, Asokkumar R, Adler DG. Clinical efficacy of gastric per-oral endoscopic myotomy (G-POEM) in the treatment of refractory gastroparesis and predictors of outcomes: a systematic review and meta-analysis using surgical pyloroplasty as a comparator group. Surg Endosc. 2020 Aug;34(8):3352-3367. doi: 10.1007/s00464-019-07135-9. Epub 2019 Oct 3. PMID 31583465
- See also: Safety information for TransPyloric Shuttle/TransPyloric Shuttle Delivery Device — https://www.accessdata.fda.gov/cdrh_docs/pdf18/P180024B.pdf